CLINICAL TRIAL: NCT03389958
Title: Safe Maternity Care Through Immediate Provision of Highly-effective Postpartum Contraception
Brief Title: Maternity Care and Contraception
Acronym: COMSE
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: Universidad de Antioquia (Other)
Responsible Party: Principal Investigator, Maureen Baldwin, Assistant Professor, Oregon Health and Science University
Other Study IDs: 11331
Record Dates: First submitted 2017-12-20; First posted 2018-01-04 (Actual); Last update posted 2018-01-04 (Actual); Status verified 2017-12

CONDITIONS: Contraception; Maternal Care Patterns; Pregnancy Related
Keywords: intrauterine device; postpartum contraception; repeat pregnancy; adolescent pregnancy
MeSH Terms: interventions — Counseling

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Counseling and provision of contraception — Provider training, availability of contraceptive methods
  Other Names: Copper IUD, Jadelle

SUMMARY:
This is a multicenter observational study of implementation of postpartum contraceptive counseling and provision into the maternity care setting in Colombia, South America. The primary aim is to determine proportion of uptake of highly-effective contraceptive use after these methods become available immediately postpartum. Secondary aims include rapid repeat pregnancy rates, use of other types of contraception, breastfeeding continuation, and visualization of IUD strings after immediate postpartum placement.

DETAILED DESCRIPTION:
This pre- post-intervention study will take place in Colombia, South America in 2 cities: Medellin (2 sites and Cartagena 1 site). The main objective is to determine the proportion of contraceptive usage by women who have just had a baby, before and after the introduction of specialized contraceptive counseling into maternity care and availability of the most effective contraceptive methods:

Group 1 (Standard of care) participants will be asked about intention for contraception usage upon hospital discharge after maternity care.

Group 2 (Intervention) participants will receive standardized contraceptive counseling and immediate access to the method of choice, including long acting reversible contraception (LARC) and other locally available methods. LARC methods available in Colombia include the copper-T intrauterine device (IUD) and Jadelle® implant, both of which are safe for usage in postpartum women.

Both groups will undergo follow- up via phone at 6-8 weeks, and 6 and 12 months postpartum to determine contraceptive continuation, repeat pregnancy, and to track any complications with the usage of LARC, including infection and contraceptive failure. For subjects with an IUD, an additional visit would take place at 8-10 days to determine need for IUD string trimming and visualization of strings.

The intervention will include introduction of specialized standardized contraceptive counseling to occur during inpatient maternity care and immediate postpartum availability of LARC methods. Currently, contraceptive counseling is left to the postpartum primary care setting and obstetric providers are not trained for immediate IUD placement. LARC devices are not typically available in the inpatient setting. Providers and staff of all levels will be trained in standardized contraceptive counseling methods. Obstetric providers will be trained in immediate postplacental IUD insertion. Staff nurses and providers will have access to company-sponsored implant insertion training programs.

The proportion of participants using LARC methods after implementation of the intervention will be compared to the proportion choosing LARC prior to the intervention. Additionally, the outcomes of women choosing non-LARC methods will be compared to those choosing LARC methods.

The study has received funding by the Colombian grant agency, Colciencias. Regulatory oversight has previously been granted by the University of Antioquia's (Medellin, Colombia) Institutional Review Board. Research operations are managed by the local Colombian organization, NACER, with support of research design and methods, statistical analysis, and medical expertise and trainings provided by clinicians from OHSU. Day to day research operations will be managed by research coordinators at each of the three maternity care hospital sites with support and monitoring by NACER and by OHSU clinicians.

The role of OHSU clinicians will be to provide research infrastructure and clinical support via remote communications, to provide initial training of trainers, to provide monitoring of recruitment and counseling methods, to help in the creation and monitor quality of data collection forms, and to perform statistical analyses. OHSU will not participate in recruitment of participants or in clinical procedures. We do not plan to be present at any research sites in person, though may perform monitoring visits if funds are available.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman in labor
* Live fetus over 20 weeks gestation
* Age >14 years

Exclusion Criteria:

* No medical exclusions for the contraceptive method chosen

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women undergoing management of a pregnancy that results in live birth over 20 weeks gestation during the same hospitalization at three public hospitals in Colombia (in Cartagena and Medellin).
Sampling Method: Non-Probability Sample
Enrollment: 299 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2016-12-30 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Proportion of women receiving immediate postpartum long-acting contraception | Through hospital discharge (an average of 3 days)
  The proportion of women who receive immediate long-acting contraception prior to hospital discharge following the intervention phase of training and availability of devices will be compared to a baseline group prior to the implementation.

SECONDARY OUTCOMES:
Continuation of long-acting contraception placed immediately postpartum | 6, 12 and 18 months postpartum
  Phone followup will be used to determine the proportion of women who are continuing their contraceptive method
Complications of contraception | 6, 12 and 18 months postpartum
  Phone followup will be used to determine the proportion of women who have experienced any complications from contraception
Comparison of long-acting methods to short-acting methods | 6, 12, and 18 months postpartum
  Outcomes (pregnancy, discontinuation) of women choosing long-acting methods will be compared to short-acting methods, coital dependent methods, or no method

CONTACTS AND LOCATIONS:
Locations (3):
- Colombia (3):
  - Maternidad Rafael Calvo, Cartagena
  - Hospital General de Medellin, Medellín
  - Metrosalud Manrique, Medellín

IPD SHARING:
Plan to Share IPD: No